CLINICAL TRIAL: NCT04366934
Title: Study of the Pathogenesis of Olfactory Disorders in COVID-19
Acronym: COVIDSMELL
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Hôpital Lariboisière, AP-HP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-021
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Coronavirus Infection; Severe Acute Respiratory Syndrome; Sars-CoV2
Keywords: SARS-CoV-2; Sense of smell disorders; Anosmia; Olfaction; Nasal neuroepithelium; Olfactory mucosa
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; Anosmia | interventions — Taste

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients: Subject consulting in the Lariboisière hospital (Paris) in the context of the COVID-19 screening care for a suspected SARS-CoV-2 infection
  Interventions: Other: Nasal swab; Other: Taste and olfactory function evaluation
- Control subjects: Subject consulting in the ear, nose and throat department at the Lariboisière hospital (Paris) with no biologically confirmed COVID-19 or suspected COVID-19 in the past 8 weeks, and no symptoms suggestive of COVID-19 or another respiratory disease and therefore no recent anosmia or ageusia
  Interventions: Other: Nasal swab; Other: Taste and olfactory function evaluation

INTERVENTIONS:
Other: Nasal swab — Nasal swab
Other: Taste and olfactory function evaluation — Taste and olfactory function evaluation

SUMMARY:
This study is a case-control study to characterize the molecular and cellular anomalies of the olfactory epithelium of COVID-19 patients with isolated anosmia, by comparison with the olfactory epithelium of non-infected subjects.

DETAILED DESCRIPTION:
Olfactory and taste dysfunctions are common and early onset in COVID-19, especially in pauci symptomatic patients, and may be the main clinical manifestations of the infection. Olfactory dysfunction could result from infection of the olfactory system by SARS-CoV-2 or from inflammation induced by the virus. While the recent development of COVID-19 pulmonary lesion research has revealed a viral, inflammatory and vascular origin, factors that cause olfactory disorders in COVID-19 are just beginning.

Acute anosmia observed in some patients with COVID-19 could result from:

* the direct infection of olfactory sensory neurons or neural stem cells of the olfactory mucosa,
* an underlying inflammation of the olfactory mucosa, leading to possible neurodegeneration of olfactory sensory neurons, and neural stem cells of the olfactory mucosa, by analogy with the respiratory viruses responsible for chronic rhinosinusitis.

It is therefore necessary to conduct a virological, cellular, immunological and inflammatory study of the olfactory epithelium from COVID-19 patients with isolated anosmia to identify the origin of these olfactory disorders.

This study is a case-control study to characterize the molecular and cellular anomalies of the olfactory epithelium of COVID-19 patients with isolated anosmia, by comparison with the olfactory epithelium of non-infected subjects.

Following measures will be performed at inclusion :

* Taste and olfactory function evaluation by a self-questionnaire taste and smell survey (TTS) and a visual analogue scale (VAS)
* Nasal swab sampling for collection of epithelium cells and olfactory mucus.

ELIGIBILITY:
Inclusion Criteria:

COVID-19 patients

* Age > 18 years
* Subject consulting in the context of the COVID-19 screening care for a suspected SARS-CoV-2 infection

Controls

* Age > 18 years
* Subject consulting in the ear, nose and throat department with no biologically confirmed COVID-19 or suspected COVID-19 in the past 8 weeks, and no symptoms suggestive of COVID-19 or another respiratory disease and therefore no recent anosmia or ageusia

Exclusion Criteria (both COVID-19 patients and controls):

* Refusal or contraindication to nasal swab
* Presence of nasal sinus pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients and control subjects
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Molecular and cellular defects in olfactory epithelium | 30 months
  Ratio of olfactory sensory cells in the nasal cytological sample

SECONDARY OUTCOMES:
Biological mechanisms involved in the pathogenesis of the disease | 30 months
  Multiple measurements will be analyzed to characterize the immune and inflamatory status of the olfactory mucosa (presence of infiltrated immune cells, activation state of the immune cells in the epithelium, cytokine and interleukin level)
Epidemiological characteristics | 30 months
  Demographic variables (sex, age, blood type), risk factors (tobacco, overweight, diabetes, rhinosinusitis disease, respiratory allergy)
Olfactory and taste dysfunction | 30 months
  Self-questionnaire taste and smell survey (TTS)
Olfactory and taste dysfunction | 30 months
  Visual analogue scale (VAS) (units from 0 normal perception to 100 no perception)

CONTACTS AND LOCATIONS:
Overall Officials: Françoise LAZARINI, PhD, Study Director — Institut Pasteur
Locations (2):
- France (2):
  - Hôpital Lariboisière, Policlinique, Paris
  - Hôpital Lariboisière, Service ORL, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Melo GD, Lazarini F, Levallois S, Hautefort C, Michel V, Larrous F, Verillaud B, Aparicio C, Wagner S, Gheusi G, Kergoat L, Kornobis E, Donati F, Cokelaer T, Hervochon R, Madec Y, Roze E, Salmon D, Bourhy H, Lecuit M, Lledo PM. COVID-19-related anosmia is associated with viral persistence and inflammation in human olfactory epithelium and brain infection in hamsters. Sci Transl Med. 2021 Jun 2;13(596):eabf8396. doi: 10.1126/scitranslmed.abf8396. Epub 2021 May 3. PMID 33941622